CLINICAL TRIAL: NCT02556372
Title: A Phase 2, Pilot Study of JKB-122 to Assess Liver Tests (ALT) in Autoimmune Hepatitis (AIH) Patients Who Are Refractory or Intolerant to Current Therapies
Brief Title: Liver Test Study of Using JKB-122 in Autoimmune Hepatitis (AIH) Patients Who Are Refractory or Intolerant to Current Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiwanJ Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JKB-122AIH
Record Dates: First submitted 2015-09-20; First posted 2015-09-22 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Autoimmune Hepatitis
Keywords: AIH; JKB-122; autoimmune; hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune; Hepatitis | interventions — JKB-122

STUDY DESIGN:
Intervention Model Description: The patient takes 5mg up to 40mg depending on the monthly response.
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JKB-122 (Experimental): AIH-positive subjects (n=20) who are intolerant, refractory, ineligible or unwilling to take current therapies, and have liver enzymes that are 2 to 10 times the upper limit of normal
  Interventions: Drug: JKB-122

INTERVENTIONS:
Drug: JKB-122 — Orally administered capsules of JKB-122 which will be taken once daily with dose escalation from 5mg up to 40mg depending on the monthly response.

SUMMARY:
This is a Phase 2, pilot study in which JKB-122 is given once daily for 24 weeks in subjects with autoimmune hepatitis (AIH) who have liver enzymes that are 1.25 to 10 times the upper limit of normal (ULN) and who have had a failed response to, incomplete response to, intolerant to, ineligible to, or unwilling to take current immunosuppressant therapies. The dose of JKB-122 will be escalated monthly.

DETAILED DESCRIPTION:
This is a Phase 2, pilot study in which JKB-122 is given once daily for 24 weeks to subjects with AIH who have liver enzymes that are 1.25 to 10 times the upper limit of normal (ULN) and who have had a failed response to, incomplete response to, intolerant to, ineligible to or unwilling to take current immunosuppressant therapies. Current immunosuppressant therapy is defined as prednisone or other steroids with or without azathioprine. Failed response is defined as being non-responsive to or worsening in symptoms (elevated Alanine Aminotransferase (ALT)/aspartate aminotransferase (AST) and/or total bilirubin) despite compliance with the standard of care (SOC) over a 6 months period. Incomplete response is defined as lack of a sustained normalization of elevated ALT/AST to current standard of care (SOC) for at least 6 months. "Refractory" to the current therapy includes patients who had a failed response to, or incomplete response to the current therapy.

Subjects will be at least 18 years of age, either male or female and will have been on therapy for AIH and have not had a normalization of ALT with the current therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has definite or probable AIH diagnosis.
* Has had a liver biopsy or Fibroscan™ within 3 years and the severity of hepatic dysfunction is limited to the following:

  * Metavir Stage 0 to stage 3 fibrosis (according to liver biopsy) or Fibroscan™ results
  * ALT and AST values not exceeding 10x ULN
  * Normal bilirubin and prothrombin time (PT/INR)
* Has elevated liver test results (ALT) at least 1.25 x ULN and not exceeding 10 x ULN at baseline.
* Has had a failed response, incomplete response, intolerant, ineligible or unwilling to take current immunosuppressive therapies. Current immunosuppressive therapy is defined as prednisone or other steroids with or without azathioprine.

Exclusion Criteria:

* Has history of allergy to JKB-122 or related compounds
* Has human immunodeficiency virus (HIV) or is hepatitis B virus or hepatitis C virus (HCV) positive
* Has positive urine drug screen at Screening
* Has been diagnosed with other overlapping liver diseases such as primary biliary cirrhosis (PBC) or primary sclerosing cholangitis (PSC)
* Is currently consuming alcoholic drinks greater than 25g/day and within 3 months prior to the first screening visit.
* Is being treated with any prescription narcotic drug (including transdermal delivery systems)
* Concurrent medications within 30 days prior to screening:

  * Opioids
  * Thioridazine
  * Silymarin and related medications
  * Potentially hepatotoxic drugs
* Has a known or suspected central nervous system disorder that may predispose to seizures or lower the seizure threshold
* Has unstable and uncontrollable hypertension (>180/110 mmHg) or a blood pressure reading at baseline of 150/90 mmHg on 2 occasions separated by a 30 minute interval
* Is currently receiving dietary supplements other than a multivitamin to treat AIH
* Has received other investigational agents within 90 days prior to the first screening visit
* Has impaired renal function
* Has malignancy.
* If female, pregnant or lactating
* Has history of gastroesophageal varices, ascites, hepatic encephalopathy, hepatocellular carcinoma, and s/p liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Changes in ALT in AIH subjects given daily doses of JKB-122 | baseline and 24 weeks
  To assess changes in ALT in AIH subjects given daily doses of JKB-122

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chu Shih, PhD, Study Director — TaiwanJ Pharmaceuticals
Locations (16):
- United States (16):
  - Ruane Clinical Research Group, Inc., Los Angeles, California
  - University of California Davis Medical Center - Ticon 1, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Tulane University, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - Advanced Liver Therapies, Baylor College of Medicine, Houston, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Taxes Liver Institute, San Antonio, Texas
  - Swedish Medical Center - Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Chung YY, Rahim MN, Heneghan MA. Autoimmune hepatitis and pregnancy: considerations for the clinician. Expert Rev Clin Immunol. 2022 Apr;18(4):325-333. doi: 10.1080/1744666X.2022.2044307. Epub 2022 Mar 2. PMID 35179437